CLINICAL TRIAL: NCT00611481
Title: Phase II Study of Tai Chi Exercise in Relation to Balance in Persons With Parkinson's Disease
Brief Title: Study of Tai Chi Exercise and Balance in Persons With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS047130 (NIH); R01NS047130 (NIH); NS047130
Record Dates: First submitted 2008-02-06; First posted 2008-02-11 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tai Ji; Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tai Chi (Experimental)
  Interventions: Behavioral: Tai Chi
- B. Strength training (Active Comparator)
  Interventions: Behavioral: Strength training
- C. Low-Impact (Other)
  Interventions: Behavioral: Low-Impact Exercise Control

INTERVENTIONS:
Behavioral: Tai Chi — a set of pre-designed Tai Chi Movements
  Arms: Tai Chi
Behavioral: Strength training — Lower-extremity strength training exercises
  Arms: B. Strength training
Behavioral: Low-Impact Exercise Control — a set of chair-based low-impact exercises
  Arms: C. Low-Impact

SUMMARY:
Patients practicing Tai Chi will exhibit significant improvements in primary outcome measures of balance, and secondary outcomes of gait, physical performance, Unified Parkinson's Disease Rating Scale, Falls, muscle strength.

DETAILED DESCRIPTION:
The study is designed to determine the effects of Tai Chi training on balance and other functional outcomes in persons with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

Patients who have:

* A diagnosis of idiopathic PD, with a disease severity rating of stage I to IV on the Hoehn and Yahr scale (Hoehn & Yahr, 1967)
* At least 1 score of 2 or more for at least 1 limb for either the tremor, rigidity, or bradykinesia item of the Unified Parkinson's Disease Rating Scale (UPDRS)
* Stable medication usage
* Not participated in a structured exercise program (i.e., not involved in any routine, organized physical activity program lasting 30 minutes or more per day, such as a gym program or regularly scheduled instructor-led exercise class) in the previous 2 months
* Ability to stand unaided or walk independently; had a personal physician's or neurologist's clearance for participation; and had a willingness to be assigned to intervention conditions.

Exclusion Criteria:

Patients who:

* Participate in any other behavioral or pharmacological research study
* Have cognitive decline (Mini-Mental State Examination score, ≤ 24) (Folstein et al., 1975)
* Have self-reported diagnosis of Alzheimer disease or other severe neurological (stage III and IV PD)
* Have evidence of progressive or debilitating conditions (metastatic cancer, severe heart or lung disease, crippling arthritis) or severe losses in vision and hearing that would limit their tolerance to testing and training procedures, that would interfere with study participation
* Are unavailable during the study period.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Balance | 3 time points

SECONDARY OUTCOMES:
gait, physical performance, Unified Parkinson's Disease Rating Scale, falls, Muscle strength | 3 time points

CONTACTS AND LOCATIONS:
Overall Officials: Fuzhong Li, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Li F, Harmer P. Economic Evaluation of a Tai Ji Quan Intervention to Reduce Falls in People With Parkinson Disease, Oregon, 2008-2011. Prev Chronic Dis. 2015 Jul 30;12:E120. doi: 10.5888/pcd12.140413. PMID 26226067
- [Derived] Li F, Harmer P, Fitzgerald K, Eckstrom E, Stock R, Galver J, Maddalozzo G, Batya SS. Tai chi and postural stability in patients with Parkinson's disease. N Engl J Med. 2012 Feb 9;366(6):511-9. doi: 10.1056/NEJMoa1107911. PMID 22316445